CLINICAL TRIAL: NCT03887455
Title: A Placebo-Controlled, Double-Blind, Parallel-Group, 18-Month Study With an Open-Label Extension Phase to Confirm Safety and Efficacy of BAN2401 in Subjects With Early Alzheimer's Disease
Brief Title: A Study to Confirm Safety and Efficacy of Lecanemab in Participants With Early Alzheimer's Disease
Acronym: Clarity AD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAN2401-G000-301; 2018-004739-58 (EudraCT Number)
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Early Alzheimer's Disease
Keywords: BAN2401; Clinical Dementia Rating-Sum of Boxes; Mild cognitive impairment; Alzheimer's disease/prodromal Alzheimer's disease; Mild Alzheimer's disease dementia; Clarity AD; Lecanemab
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — lecanemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Core Study: Lecanemab 10 mg/kg biweekly (Experimental)
  Interventions: Drug: Lecanemab IV
- Core Study: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Extension Phase: Lecanemab 10 mg/kg biweekly (Experimental)
  Interventions: Drug: Lecanemab IV
- Extension Phase: Lecanemab Subcutaneous Injection Dose 1 (Experimental): This will include approximately 40 de novo participants (those that did not participate in the core study) with early Alzheimer disease (AD).
  Interventions: Drug: Lecanemab SC
- Extension Phase: Lecanemab Subcutaneous Injection Dose 2 (Experimental)
  Interventions: Drug: Lecanemab SC
- Extension Phase: Lecanemab Subcutaneous Injection Dose 3 (Experimental)
  Interventions: Drug: Lecanemab SC
- Extension Phase: Lecanemab Subcutaneous Injection Dose 4 (Experimental)
  Interventions: Drug: Lecanemab SC
- Extension Phase: Lecanemab 10 mg/kg Intravenous Infusion Once Every 4 Weeks (Experimental)
  Interventions: Drug: Lecanemab IV
- Extension Phase B (Experimental): Participants will receive Lecanemab 10 mg/kg intravenous infusion once every 2 weeks, or 4 weeks, or Dose 3, or Dose 4 subcutaneous injection weekly.
  Interventions: Drug: Lecanemab IV; Drug: Lecanemab SC

INTERVENTIONS:
Drug: Lecanemab IV — Administered as IV infusion.
  Other Names: BAN2401
  Arms: Core Study: Lecanemab 10 mg/kg biweekly; Extension Phase B; Extension Phase: Lecanemab 10 mg/kg Intravenous Infusion Once Every 4 Weeks; Extension Phase: Lecanemab 10 mg/kg biweekly
Drug: Placebo — Biweekly (once every 2 weeks) administered as intravenous infusion.
  Arms: Core Study: Placebo
Drug: Lecanemab SC — Administered weekly as a subcutaneous injection.
  Other Names: BAN2401
  Arms: Extension Phase B; Extension Phase: Lecanemab Subcutaneous Injection Dose 1; Extension Phase: Lecanemab Subcutaneous Injection Dose 2; Extension Phase: Lecanemab Subcutaneous Injection Dose 3; Extension Phase: Lecanemab Subcutaneous Injection Dose 4

SUMMARY:
This study will be conducted to evaluate the efficacy of lecanemab in participants with early Alzheimer's disease (EAD) by determining the superiority of lecanemab compared with placebo on the change from baseline in the Clinical Dementia Rating-Sum of Boxes (CDR-SB) at 18 months of treatment in the Core Study. This study will also evaluate the long-term safety and tolerability of lecanemab in participants with EAD in the Extension Phase and whether the long-term effects of lecanemab as measured by the CDR-SB at the end of the Core Study is maintained over time in the Extension Phase. Extension Phase Part B will continue dosing with lecanemab in countries where lecanemab may not be commercially available.

DETAILED DESCRIPTION:
All administrations of study drug will be administered in the clinic or in the home; However, home administrations of intravenous (IV) study drug will be allowed per sponsor approval according to country and local guidelines during the COVID-19 pandemic and following its resolution, where permitted.

ELIGIBILITY:
Core Study: Inclusion Criteria

Diagnosis: Mild Cognitive Impairment (MCI) due to Alzheimer's disease - intermediate likelihood:

* Meet the National Institute of Aging - Alzheimer's Association (NIA-AA) core clinical criteria for MCI due to Alzheimer's disease - intermediate likelihood
* Have a global Clinical Dementia Rating (CDR) score of 0.5 and CDR Memory Box score of 0.5 or greater at Screening and Baseline
* Report a history of subjective memory decline with gradual onset and slow progression over the last 1 year before Screening; must be corroborated by an informant

Mild Alzheimer's disease dementia:

* Meet the NIA-AA core clinical criteria for probable Alzheimer's disease dementia
* Have a global CDR score of 0.5 to 1.0 and a CDR Memory Box score of 0.5 or greater at Screening and Baseline

Key Inclusion Criteria that must be met by all participants:

* Objective impairment in episodic memory as indicated by at least 1 standard deviation below age-adjusted mean in the Wechsler Memory Scale IV-Logical Memory (subscale) II (WMS-IV LMII)
* Positive biomarker for brain amyloid pathology
* Male or female participants aged greater than or equal to (>=) 50 and less than or equal to (<=) 90 years, at the time of informed consent
* Mini mental state examination (MMSE) score >=22 at Screening and Baseline and <=30 at Screening and Baseline
* Body mass index (BMI) greater than (>)17 and less than (<) 35 at Screening
* If receiving an approved Alzheimer's disease treatment such as acetylcholinesterase inhibitor (AChEIs) or memantine or both for Alzheimer's disease, must be on a stable dose for at least 12 weeks prior to Baseline. Treatment-naive participants for Alzheimer's disease can be entered into the study. Unless otherwise stated, participants must have been on stable doses of all other (that is, non-Alzheimer's disease-related) permitted concomitant medications for at least 4 weeks prior to Baseline. Use of memantine will not be allowed for participants in Japan
* Have an identified study partner (defined as a person able to support the participant for the duration of the study and who spends at least 8 hours per week with the participant)
* Provide written informed consent. If a participant lacks capacity to consent in the investigator's opinion, the participant's assent should be obtained, if required in accordance with local laws, regulations and customs, plus the written informed consent of a legal representative should be obtained (capacity to consent and definition of legal representative should be determined in accordance with applicable local laws and regulations). In countries where local laws, regulations, and customs do not permit participants who lack capacity to consent to participate in this study (example, Germany and Spain), they will not be enrolled

Extension Phase: Inclusion Criteria:

* Participants who have completed the Core Study (except de novo participants)
* Must continue to have a study partner who is willing and able to provide follow-up information on the participant throughout the course of the Extension Phase
* Provide written informed consent for the Extension Phase. If a participant lacks capacity to consent in the investigator's opinion, the participant's assent should be obtained, if required and in accordance with local laws, regulations and customs, plus the written informed consent of a legal representative should be obtained (capacity to consent and definition of legal representative should be determined in accordance with applicable local laws and regulations). In countries where local laws, regulations, and customs do not permit participants who lack capacity to consent to participate in this study (example, Germany and Spain), they will not be enrolled
* Participants entering the subcutaneous (vial) substudy at Extension Phase Week 1, must be willing to participate, or continue participating in the amyloid positron emission tomography (PET) substudy. All participants must have an amyloid PET scan within 4 weeks before starting subcutaneous BAN2401
* Participants enrolling into the subcutaneous autoinjector substudy must have had at least 6 months exposure to BAN2401 10 mg/kg intravenously biweekly or BAN2401 Dose 1 subcutaneously weekly.
* Participants enrolling into the subcutaneous Dose 3 autoinjector substudy must have previously received BAN2401 by either intravenous administration and/or subcutaneous autoinjector administration and must have completed Visit 82 (Extension Week 79) at a minimum, regardless of previous route of administration

Extension Phase Part B: Inclusion Criteria:

• Must have completed Week 207 in the Extension Phase

Exclusion Criteria

* Any neurological condition that may be contributing to cognitive impairment above and beyond that caused by the participant's Alzheimer's disease
* History of transient ischemic attacks (TIA), stroke, or seizures within 12 months of Screening
* Any psychiatric diagnosis or symptoms (example, hallucinations, major depression, or delusions) that could interfere with study procedures in the participant
* Geriatric Depression Scale (GDS) score >=8 at Screening
* Contraindications to MRI scanning, including cardiac pacemaker/defibrillator, ferromagnetic metal implants (example in skull and cardiac devices other than those approved as safe for use in MRI scanners)
* Evidence of other clinically significant lesions on brain MRI at Screening that could indicate a dementia diagnosis other than Alzheimer's disease
* Other significant pathological findings on brain MRI at screening, including but not limited to: more than 4 microhemorrhages (defined as 10 millimeter [mm] or less at the greatest diameter); a single macrohemorrhage >10 mm at greatest diameter; an area of superficial siderosis; evidence of vasogenic edema; evidence of cerebral contusion, encephalomalacia, aneurysms, vascular malformations, or infective lesions; evidence of multiple lacunar infarcts or stroke involving a major vascular territory, severe small vessel, or white matter disease; space occupying lesions; or brain tumors (however, lesions diagnosed as meningiomas or arachnoid cysts and <1 centimeter [cm] at their greatest diameter need not be exclusionary)
* Any immunological disease which is not adequately controlled, or which requires treatment with immunoglobulins, systemic monoclonal antibodies (or derivatives of monoclonal antibodies), systemic immunosuppressants, or plasmapheresis during the study
* Participants with a bleeding disorder that is not under adequate control (including a platelet count <50,000 or international normalized ratio [INR] >1.5 for participants who are not on anticoagulant treatment, example, warfarin). Participants who are on anticoagulant therapy should have their anticoagulant status optimized and be on a stable dose for 4 weeks before Screening. Participants who are on anticoagulant therapy are not permitted to participate in cerebrospinal fluid (CSF) assessments
* Any other medical conditions (example, cardiac, respiratory, gastrointestinal, renal disease) which are not stably and adequately controlled, or which in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
* Participation in a clinical study involving any therapeutic monoclonal antibody, protein derived from a monoclonal antibody, immunoglobulin therapy, or vaccine within 6 months before screening unless it can be documented that the participant was randomized to placebo
* Participation in a clinical study involving any anti-amyloid therapies (including any monoclonal antibody therapies and any β-site amyloid precursor protein cleaving enzyme [BACE] inhibitor therapies) unless it can be documented that the participant only received placebo
* Participants who have any known prior exposure to lecanemab
* Participants who were dosed in a clinical study involving any new chemical entities for AD within 6 months prior to screening unless it can be documented that the participant was in a placebo treatment arm

Extension Phase: Exclusion Criteria

* Participants who discontinued early from the Core Study
* Participants who develop the following conditions from the time of Screening for the Core Study to the start of the Extension Phase

  * Any neurological condition that may be contributing to cognitive impairment above and beyond that caused by the participant's AD
  * Any psychiatric diagnosis or symptoms, (example, hallucinations, major depression, or delusions) that could interfere with study procedures in the participant
  * Contraindications to MRI scanning, including cardiac pacemaker/defibrillator, ferromagnetic metal implants (example, in skull and cardiac devices other than those approved as safe for use in MRI scanners)
  * Other significant pathological findings on brain MRI during the Core Study including but not limited to: cerebral contusion, encephalomalacia, aneurysms, vascular malformations, or infective lesions; evidence of multiple lacunar infarcts or stroke involving a major vascular territory, severe small vessel, or white matter disease; space occupying lesions; or brain tumors will be exclusionary if based on the opinion of the investigator, with consultation of medical monitor, these findings may interfere with the study procedures or safety
  * Hypersensitivity to BAN2401 or any of the excipients, or to any monoclonal antibody treatment
  * Any immunological disease which is not adequately controlled, or which requires chronic treatment with immunoglobulins, systemic monoclonal antibodies (or derivatives of monoclonal antibodies), systemic immunosuppressants, or plasmapheresis during the study
  * Any other clinically significant abnormalities in physical examination, vital signs, laboratory tests, or ECG, which in the opinion of the investigator require further investigation or treatment or which may interfere with study procedures or safety
  * Malignant neoplasms (except for basal or squamous cell carcinoma in situ of the skin, or localized prostate cancer in male participants) that are not stably and adequately controlled or which, based on the opinion of the investigator, may interfere with the participant's safety or participation in the study
  * Any other medical conditions (example, cardiac, respiratory, gastrointestinal, renal disease) which are not stably and adequately controlled, or which in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
  * Severe visual or hearing impairment that would prevent the participant from performing psychometric tests accurately

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1906 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Core Study: Change from Baseline in the CDR-SB at 18 Months | Baseline, 18 months
Extension Phase: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) | From first dose of study drug up to approximately 51 months (including 3 months follow up) for the extension phase
  A TEAE is defined as an adverse event that emerges during treatment or within 30 days of the last dose of study drug, having been absent at pretreatment (Baseline) or reemerges during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or worsens in severity during treatment relative to the pretreatment state, when the adverse event was continuous. Number of participants with TEAEs (serious and non-serious adverse events) will be reported based on their regular measurement of vital signs, safety assessments of laboratory tests, antidrug antibody assessments, suicidality assessments, magnetic resonance imaging and electrocardiogram parameter values.
Extension Phase: Change from Core Study Baseline in CDR-SB | Baseline up to Month 66
Extension Phase Part B: Number of Participants Exposed to Lecanemab | From 48th month in extension phase part A to the end of extension phase part B (up to 24 months)

SECONDARY OUTCOMES:
Core Phase: Change From Baseline in Amyloid Positron Emission Tomography (PET) Using Centiloids at 18 Months | Baseline, 18 months
Core Study: Change from Baseline in Alzheimer Disease Assessment Scale - Cognitive Subscale 14 (ADAS-cog14) at 18 Months | Baseline, 18 months
Core Phase: Change From Baseline in Alzheimer's Disease Composite Score (ADCOMS) at 18 Months | Baseline, 18 months
Core Study: Change From Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living Scale for Mild Cognitive Impairment (ADCS MCI-ADL) at 18 Months | Baseline, 18 months
Extension Phase Part B: Number of Participants Reporting Adverse Events | From 48th month in extension phase part A to the end of extension phase part B (up to 24 months)

CONTACTS AND LOCATIONS:
Locations (246):
- United States (111):
  - Banner Alzheimer's Institute- Clinical Trials Department, Phoenix, Arizona
  - Banner Sun Health Research, Sun City, Arizona
  - Neurological Associates of Tucson dba Center for Neurosciences, Tucson, Arizona
  - Neurology Center of North Orange County, Fullerton, California
  - Irvine Clinical Research, Irvine, California
  - University of California - Los Angeles, Los Angeles, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - Stanford University Medical Center, Palo Alto, California
  - Pacific Research Network, Inc, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - UCSF Memory and Aging Center, San Francisco, California
  - Apex Research Institute, Santa Ana, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - North Bay Neuroscience Research Institute, Sebastopol, California
  - ImmunoE Research Center, Centennial, Colorado
  - Mile High Research Center, Denver, Colorado
  - Associated Neurologists of Southern Connecticut, Fairfield, Connecticut
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Yale University School Of Medicine, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - JEM Research Institute, Atlantis, Florida
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Advanced Clinical Research Network, Coral Gables, Florida
  - Linfritz Research Institute, Inc., Coral Gables, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest FL, Fort Myers, Florida
  - Infinity Clinical Research, Hollywood, Florida
  - Charter Research, Lady Lake, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Clincloud, LLC, Maitland, Florida
  - Gonzalez MD & Aswad MD Health Services, Miami, Florida
  - BioMed Research Institute, Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - CCM Clinical Research Group, Miami, Florida
  - Rios Medical Center, Inc., Miami, Florida
  - Vitae Research Center, Miami, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Visionary Investigators Network, Miami, Florida
  - Allied Biomedical Research (Clinical Trial), Miami, Florida
  - Pharmax Research of South Florida, Inc, Miami, Florida
  - Galiz Research, Miami Springs, Florida
  - Renstar Medical Research, Ocala, Florida
  - Bioclinica Research, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Advanced Research Consultants, Inc., Palm Beach Gardens, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Quantum Laboratories Inc., Pompano Beach, Florida
  - Neurostudies, Inc., Port Charlotte, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Alzheimer's Research and Treatment Center, Stuart, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - USF Suncoast Gerontology Center, Tampa, Florida
  - Bioclinica Research, The Villages, Florida
  - Premiere Research Institute, West Palm, West Palm Beach, Florida
  - Emory University Cognitive Neurology Clinic & ADRC, Atlanta, Georgia
  - Columbus Memory Center, Columbus, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - NeuroStudies.net, LLC, Decatur, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - KU Wichita Center for Clinical Research, Wichita, Kansas
  - Partners Population Health, Belmont, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - ActivMed Practices & Research, Methuen, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Donald S. Marks, MD. P.C., Plymouth, Massachusetts
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Washington University, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Advanced Memory Research Institute of NJ, PC, Toms River, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Albany Medical College, Albany, New York
  - Neurological Associates of Albany, PC, Albany, New York
  - New York University Medical Center PRIME, New York, New York
  - Neurological Institute of New York, New York, New York
  - University of Rochester, Rochester, New York
  - ANI Neurology, PLLC d/b/a Alzheimer's Memory Center, Charlotte, North Carolina
  - Raleigh Neurology Associates, P.A. - Research Department, Raleigh, North Carolina
  - PMG Research of Winston Salem, Winston-Salem, North Carolina
  - OH Clinical Research Partners, Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Columbs Neuroscience, LLC, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Summit Research Network (OR) Inc., Portland, Oregon
  - Neural Net Research, LLC, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital - Memory and Aging Program, Providence, Rhode Island
  - Roper St. Francis Healthcare, North Charleston, South Carolina
  - Coastal Neurology, P.A., Port Royal, South Carolina
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Alliance for Multispecialty Research LLC, New Orleans Center for Clinical Research / Volunteer Research Group, an AMR company, Knoxville, Tennessee
  - Senior Adult Specialty Research, Austin, Texas
  - Texas Neurology, PA, Dallas, Texas
  - Kerwin Research Center, Dallas, Texas
  - Baylor College of Medicine AD and Memory Disorders Center, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - DBA The Memory Clinic, Bennington, Vermont
  - National Clinical Research Inc.-Richmond, Richmond, Virginia
  - Kingfisher Cooperative LLC, Spokane, Washington
- Australia (7):
  - St Vincent's Hospital - Translational Research Centre, Darlinghurst, New South Wales
  - KaRa Institute of Neurological Diseases, Macquarie Park, New South Wales
  - The Prince Charles Hospital/Internal Medicine & Dementia Research Unit, Chermside Brisbane, Queensland
  - Central Adelaide Local Health Network, The Queen Elizabeth Hospital and the Royal Adelaide Hospital, Woodville South, Adelaid, South Australia
  - Austin Health - Medical and Cognitive Research Unit, Ivanhoe, Victoria
  - HammondCare Malvern Clinical Trials Unit, Malvern, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia
- Canada (11):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Health Research, West Vancouver, British Columbia
  - True North Clinical Research Halifax, Inc., Halifax, Nova Scotia
  - True North Clinical Research Kentville, Inc., Kentville, Nova Scotia
  - St. Joseph's HC- Parkwood Institute, London, Ontario
  - Recherches Neuro-Hippocampe, Inc., d/b/a Ottawa Memory Clinic, Ottawa, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program (Neurology Research Inc.), Toronto, Ontario
  - Recherches Neuro-Hippocampe Inc. d/b/a Clinique de la Mémoire de l'Outaouais, Gatineau, Quebec
  - MoCA Clinic and Institute/NeuroSearch Developpements Inc., Greenfield Park, Quebec
  - Q&T Research Sherbrooke Inc., Sherbrooke, Quebec
- China (21):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Sun Yat-Sent Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Guangzhou Huiai Hospital, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangzhou
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Nanjing Brain Hospital, Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Qinghai Provincial People's Hospital, Xining, Qinghai
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiaotong Universtiy School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- France (8):
  - Hôpital de Hautepierre, Strasbourg, Bas Rhin
  - Hopital de la Timone, Marseille, Cedex 05
  - Hôpital Gui de Chauliac, Montpellier, Cedex 5
  - Hopital Guillaume et RenÃ LaÃnnec, Nantes, Cedex
  - Groupe Hospitalier Pitie-Salpetriere, Paris, Cedex
  - Centre de Recherche Clinique du Gérontopôle, Toulouse, Haute Garonne
  - Hôpital Lariboisière, Paris, Paris
  - Hôpital neurologique Pierre Wertheimer, Bron
- Germany (6):
  - Eisai Trial Site #5, Günzburg, Baden-Wurttemberg
  - Eisai Trial Site #2, Mannheim, Baden-Wurttemberg
  - Eisai Trial Site #6, Berlin
  - Eisai Trial Site #1, Bielefeld
  - Eisai Trial Site #4, Erbach im Odenwald
  - Eisai Trial Site #3, München
- Italy (10):
  - Ospedale "Card. G. Panico" -, Tricase, LE
  - Fondazione Istituto G.Giglio di Cefalù, Cefalù, Palermo
  - Clinica Neurologica, IRCCS Ospedale Policlinico San Martino, Genova, Genova
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico - U.O.S.D. Malattie Neurodegenerative, Milan
  - ASST-Monza, Ospedale San Gerardo, Monza
  - Prima Clinica Neurologica, Primo Policlinico AOU "L. Vanvitelli", Napoli
  - Ospedale S. Maria della Misericordia, S. Andrea delle Fratte, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Fondazione Policlinico Agostino Gemelli - UCSC, Roma
  - Universita' Sapienza di Roma - Dipartimento di Neuroscienze Umane, Roma
- Japan (33):
  - Eisai Trial Site #4, Obu-shi, Aichi-ken
  - Eisai Trial Site #15, Chiba, Chiba
  - Eisai Trial Site #6, Yoshida-gun, Fukui
  - Eisai Trial Site #1, Fujioka-shi, Gunma
  - Eisai Trial Site #32, Ōtake, Hiroshima
  - Eisai Trial Site #30, Sapporo, Hokkaido
  - Eisai Trial Site #28, Himeji-shi, Hyōgo
  - Eisai Trial Site #19, Kobe, Hyōgo
  - Eisai Trial Site #24, Toride-shi, Ibaraki
  - Eisai Trial Site #9, Kahoku, Ishikawa-ken
  - Eisai Trial Site #7, Atsugi-shi, Kanagawa
  - Eisai Trial Site #17, Fujisawa-shi, Kanagawa
  - Eisai Trial Site #20, Kawasaki-shi, Kanagawa
  - Eisai Trial Site #2, Yokohama, Kanagawa
  - Eisai Trial Site #33, Higashimorokatagun, Miyazaki
  - Eisai Trial Site #22, Niigata, Niigata
  - Eisai Trial Site #16, Kurashiki-shi, Okayama-ken
  - Eisai Trial Site #8, Hirakata, Osaka
  - Eisai Trial Site #26, Suita-shi, Osaka
  - Eisai Trial Site #18, Saitama-shi, Saitama
  - Eisai Trial Site #31, Ōtsu, Shiga
  - Eisai Trial Site #5, Bunkyo-ku, Tokyo
  - Eisai Trial Site #29, Bunkyo-ku, Tokyo
  - Eisai Trial Site #13, Hachioji-shi, Tokyo
  - Eisai Trial Site #12, Musashino-shi, Tokyo
  - Eisai Trial Site #23, Shinagawa-ku, Tokyo
  - Eisai Trial Site #25, Shinjuku-ku, Tokyo
  - Eisai Trial Site #10, Shinjuku-ku, Tokyo
  - Eisai Trial Site #3, Yamagata, Yamagata
  - Eisai Trial Site #21, Hōfu, Yamaguchi
  - Eisai Trial Site #14, Ube-shi, Yamaguchi
  - Eisai Trial Site #11, Osaka
  - Eisai Trial Site #27, Osaka
- First Moscow State Medical University n.a. I.M. Sechenov, Moscow, Russia
- National University Hospital, Singapore, Singapore
- South Korea (13):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hospital, Gwangju, Jeolla-do
  - Seoul National University Bundang Hospital, Seongnam-si, Seoul
  - Dong-A University Hospital, Busan
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul
- Spain (12):
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Centro CAE Oroitu, Getxo, Bizkaia
  - Fundación CITA-alzheimer Findazioa, Donostia / San Sebastian, Gipuzkoa
  - Policlinica Guipuzcoa, Donostia / San Sebastian, Guipuzcoa
  - Fundacion ACE, Barcelona, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Santa Cruz y San Pablo, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Complejo Hospitalario Ruber Juan Bravo, Madrid
  - Hospital de Salamanca, Salamanca
  - Hospital Victoria Eugenia - Cruz Roja, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg, Västra Götalandslän
  - Memory Clinic, Malmö University Hospital, Malmo
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala, Uppsala
- United Kingdom (8):
  - Re:Cognition Health, Plymouth, Devon
  - Memory Assessment & Research Centre (MARC),, Southampton, Hampshire
  - Sheffield Memory Service, Sheffield, South Yorkshire
  - Re:Cognition Health Ltd, Birmingham
  - Re:Cognition Health Ltd, Guildford
  - St. Pancras Clinical Research, London
  - Re:Cognition Health Ltd, London
  - Charing Cross Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Devanarayan V, Ye Y, Zhu L, Tian L, Kramer L, Irizarry M, Dhadda S. Predicted natural progression as an Alzheimer's prognostic covariate improves the precision of lecanemab efficacy assessments and clinical trial efficiency. Alzheimers Dement. 2025 Mar;21(3):e70045. doi: 10.1002/alz.70045. PMID 40042496
- [Derived] Devanarayan V, Charil A, Horie K, Doherty T, Llano DA, Andreozzi E, Sachdev P, Ye Y, Murali LK, Zhou J, Reyderman L, Hampel H, Kramer LD, Dhadda S, Irizarry MC; Alzheimer's Disease Neuroimaging Initiative (ADNI). Plasma pTau217 ratio predicts continuous regional brain tau accumulation in amyloid-positive early Alzheimer's disease. Alzheimers Dement. 2025 Feb;21(2):e14411. doi: 10.1002/alz.14411. Epub 2024 Nov 22. PMID 39575854
- [Derived] Devanarayan V, Doherty T, Charil A, Sachdev P, Ye Y, Murali LK, Llano DA, Zhou J, Reyderman L, Hampel H, Kramer LD, Dhadda S, Irizarry MC. Plasma pTau217 predicts continuous brain amyloid levels in preclinical and early Alzheimer's disease. Alzheimers Dement. 2024 Aug;20(8):5617-5628. doi: 10.1002/alz.14073. Epub 2024 Jun 28. PMID 38940656
- [Derived] Honig LS, Sabbagh MN, van Dyck CH, Sperling RA, Hersch S, Matta A, Giorgi L, Gee M, Kanekiyo M, Li D, Purcell D, Dhadda S, Irizarry M, Kramer L. Updated safety results from phase 3 lecanemab study in early Alzheimer's disease. Alzheimers Res Ther. 2024 May 10;16(1):105. doi: 10.1186/s13195-024-01441-8. PMID 38730496
- [Derived] Tahami Monfared AA, Ye W, Sardesai A, Folse H, Chavan A, Aruffo E, Zhang Q. A Path to Improved Alzheimer's Care: Simulating Long-Term Health Outcomes of Lecanemab in Early Alzheimer's Disease from the CLARITY AD Trial. Neurol Ther. 2023 Jun;12(3):863-881. doi: 10.1007/s40120-023-00473-w. Epub 2023 Apr 2. PMID 37009976
- [Derived] van Dyck CH, Swanson CJ, Aisen P, Bateman RJ, Chen C, Gee M, Kanekiyo M, Li D, Reyderman L, Cohen S, Froelich L, Katayama S, Sabbagh M, Vellas B, Watson D, Dhadda S, Irizarry M, Kramer LD, Iwatsubo T. Lecanemab in Early Alzheimer's Disease. N Engl J Med. 2023 Jan 5;388(1):9-21. doi: 10.1056/NEJMoa2212948. Epub 2022 Nov 29. PMID 36449413